CLINICAL TRIAL: NCT02485353
Title: Pilot Study of Vosaroxin and Cytarabine for the Treatment of Adults 60 Years of Age or Older With Previously Untreated AML
Brief Title: Study of Vosaroxin and Cytarabine for the Treatment of Adults 60 Years of Age or Older With Previously Untreated AML
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety concerns
Sponsor: Hamid Sayar (Other)
Responsible Party: Sponsor-Investigator, Hamid Sayar, Assistant Professor of Clinical Medicine, Hematology/Oncology, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0525
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-08

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Vosaroxin; Cytarabine; Remission Induction; Safety; Progression-Free Survival; Mortality Rate; Length of Stay
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — vosaroxin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vosaroxin and Cytarabine (Other)
  Interventions: Drug: Vosaroxin and Cytarabine

INTERVENTIONS:
Drug: Vosaroxin and Cytarabine

SUMMARY:
This is a pilot efficacy assessment clinical trial of vosaroxin and cytarabine for the treatment of adults 60 years of age or older with previously untreated acute myeloid leukemia. A total of 17 evaluable patients are planned to be treated on the study.

DETAILED DESCRIPTION:
Primary objective: rate of complete remission (morphologic complete remission or morphologic complete remission with incomplete blood count recovery) Secondary objectives: (1) safety of this combination in induction therapy of older patients previously unexposed to intensive chemotherapy; (2) progression-free survival; (3) length of stay in hospital for induction; (4) 30- and 60-day mortality rate.

The treatment period will include up to 4 cycles of treatment (induction 1, induction 2, consolidation 1, and consolidation 2). In each cycle, the first day of study treatment will be considered day 1.

* Each cycle will include vosaroxin treatment on days 1 and 4 (total of 2 days) and cytarabine treatment on days 1-5 (total of 5 days) followed by a variable interval required to achieve hematologic recovery, defined as absolute neutrophil count (ANC) > 1000 cells/L.
* Up to 2 cycles of consolidation treatment may be completed by eligible patients in remission (morphologic complete remission or morphologic complete remission with incomplete blood count recovery) if safety parameters are met.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* A diagnosis of AML based on WHO classification (>20% myeloblasts in peripheral blood or bone marrow)
* No previous treatment with chemotherapy for AML, other than hydroxyurea. Previous treatment with hypomethylating agents is acceptable
* Patients must have an ECOG (Zubrod) performance status of 0-2 (see Appendix I).
* Patients must have adequate hepatic function with a total bilirubin < 1.5 times upper limit normal (ULN) other than cases of Gilbert disease, and ALT and AST < 2.5 times ULN; and adequate renal function as defined by a serum creatinine < 2 times ULN.
* Clinically significant nonhematologic toxicity after prior therapy has recovered to grade 1 per Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 or newer
* Patients must have the ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to initiation of treatment
* Left ventricular ejection fraction (LVEF) at least 40% by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)

Exclusion Criteria:

* Patients with known central nervous system (CNS) leukemia by spinal fluid cytology, flow cytometry or imaging. A lumbar puncture is not required unless CNS involvement is clinically suspected. Patients with signs or symptoms of leukemic meningitis or a history of leukemic meningitis must have a negative lumbar puncture within 2 weeks of study enrollment.
* A diagnosis of acute promyelocytic leukemia (APL). The study does not require to rule APL out for every subject. However, if there is clinical suspicion for APL, such diagnosis has to be ruled out before initiation of treatment.
* Active malignancy currently undergoing chemo or radiation therapy. Hormone therapy is acceptable.
* Active serious infection that at the discretion of treating physician makes patient ineligible for chemotherapy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Sayar, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on enrolling 20 patients. Due to the death of 2 patients which raised safety concerns, the study was closed with 2 patients enrolled.
Groups:
- Vosaroxin and Cytarabine: Each cycle will include vosaroxin treatment on days 1 and 4 (total of 2 days) and cytarabine treatment on days 1-5 (total of 5 days) followed by a variable interval required to achieve hematologic recovery, defined as absolute neutrophil count (ANC) > 1000 cells/L
Period: Overall Study
Arm/Group | Vosaroxin and Cytarabine
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vosaroxin and Cytarabine
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (1.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Remission
Description: Percentage of patients who have complete remission as defined by the International Working Group for AML: morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi or CRp)
Time Frame: 2 months
Population: All patients receiving at least one dose of study drug and having at least one evaluable post-baseline visit
Measure: Number; unit: percentage of patients
Arm/Group | Vosaroxin and Cytarabine
Number analyzed (Participants) | 2
percentage of patients | 0

2. Secondary Outcome: Procedure or Procedure Related Adverse Events
Description: Number of unique patients who had a procedure or treatment related (possible, probable or definite) adverse events. (graded per NCI CTC v4.0)
Time Frame: Up to 1 year
Population: All patients enrolled and received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vosaroxin and Cytarabine
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Vosaroxin and Cytarabine
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vosaroxin and Cytarabine (N=2)
Infections and infestations - Other (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vosaroxin and Cytarabine (N=2)
Mucositis oral (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Upper respiratory infection (Infections and infestations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Diziness (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the death of 2 patients which raised safety concerns, the study was closed with 2 patients enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes